CLINICAL TRIAL: NCT01455948
Title: Canadian Health Economics, Health Outcome, and Effectiveness Comparison of Treatment of the Frontal Sinus Ostium and Recess and Other Sinuses With Functional Endoscopic Sinus Surgery (FESS) or Balloon Sinuplasty in Patients With Chronic Sinusitis (CRS)
Brief Title: Canadian Health Economics, Outcome, and Effectiveness Comparison of Treatment in Patients With Chronic Rhinosinusitis
Acronym: CHEC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Acclarent (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: JJMC-001
Record Dates: First submitted 2011-10-11; First posted 2011-10-20 (Estimated); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Chronic Rhinosinusitis
Keywords: sinusitis; chronic; Functional endoscopic sinus surgery; balloon sinuplasty
MeSH Terms: conditions — Sinusitis; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Balloon Sinuplasty™ System (Active Comparator)
  Interventions: Device: Relieva Balloon Sinuplasty™ System
- Functional Endoscopic Sinus Surgery (Active Comparator)
  Interventions: Procedure: Functional Endoscopic Sinus Surgery

INTERVENTIONS:
Device: Relieva Balloon Sinuplasty™ System — Catheter-based devices used to dilate blocked paranasal sinus ostia (openings).
  Arms: Balloon Sinuplasty™ System
Procedure: Functional Endoscopic Sinus Surgery — Specialized probes are used to cannulate closed ostia (openings), and small forceps are used to resect periostial bone and tissue to enlarge the sinus ostia.
  Arms: Functional Endoscopic Sinus Surgery

SUMMARY:
The economic, patient related outcome, and effectiveness of balloon sinuplasty in the treatment of CRS patients with frontal and other sinus disease in the Canadian healthcare environment is not known at this time. This study will evaluate the impact of balloon sinuplasty and traditional FESS treatment on CRS patients.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of unilateral or bilateral Chronic Rhinosinusitis based on the European Position Paper on Rhinosinusitis and Nasal Polyps (2) with at least frontal and maxillary sinus involvement
* Documented failed medical treatment of CRS
* Eighteen (18) to sixty-five (65) years of age
* Employed in full time position or equivalent
* Planned FESS for treatment of CRS
* Must have an American Society of Anesthesiologists physical status of P3 classification or less
* Able to provide informed consent by signing the informed consent document at the screening visit prior to any study activities
* Able to read and understand English

Exclusion Criteria:

* Previous sinonasal surgery
* Pregnant
* Cystic Fibrosis
* Diagnosed immotile cilia syndrome
* Samter's Triad
* Diagnosed immunodeficiency syndrome
* Diagnosed fungal sinusitis
* Concurrent septoplasty or turbinate surgery
* Diagnosed recurrent acute sinusitis
* Current smoker
* Presence of grade 2 or greater nasal polyps
* Sinonasal tumors or obstructive lesions
* History of substance or alcohol abuse within the past 12 months
* Investigator's opinion that the subject should not be in the study such as any conditions that could compromise the wellbeing of the patient or integrity of the study or prevent the patient from meeting or performing study requirements
* Participation in a research study 30 days prior to surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The direct and indirect costs of treatment of frontal and other sinus disease with Functional Endoscopic Sinus Surgery or balloon sinuplasty. | 6 months

SECONDARY OUTCOMES:
Health outcome of patients in the two treatment groups. | 6 months
  Health outcomes will be determined by the completion of the EQ-5D questionnaire in both treatment groups at various timepoint. The EQ-5D is a standardised measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. Applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status that can be used in the clinical and economic evaluation of health care as well as in population health surveys.
Effectiveness of the two treatment groups in relieving symptomology of CRS. | 6 months
  Effectiveness of the two treatment groups in relieving symptomology of CRS will be determined by the completion of the Sino-nasal Outcome Test - 20 (SNOT-20) questionnaire in both treatment groups at various timepoint. The SNOT-20 questionnaire is a validated instrument for the measurement of disease specific health status and quality of life in patients with chronic rhinosinusitis.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Witterick, MD, MSc, Principal Investigator — Mount Sinai Hospital, Toronto, Ontario, Canada
Locations (8):
- Canada (8):
  - Hamilton General Hospital, Hamilton, Ontario
  - St. Joseph's Health Centre, London, Ontario
  - Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - Trillium Health Centre, Toronto, Ontario
  - Toronto East General, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario